CLINICAL TRIAL: NCT06866106
Title: The WISH Intervention for IBS: Feasibility, Preliminary Effects, and Candidate Gut-Brain Mechanisms
Brief Title: Well-being in IBS: Strengths and Happiness (WISH) 2.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth N. Madva, M.D., Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P000594
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; brain-gut behavior therapy; behavioral health intervention; psychological intervention; psychotherapy
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psychology, Positive; Methods; Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing positive psychology (PP) intervention to educational intervention
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology (PP) Intervention (Experimental): Participants will complete an adapted, optimized, phone-based, 9-week positive psychology (PP) intervention.
  Interventions: Behavioral: Positive Psychology (PP) Intervention
- Educational Intervention (Active Comparator): Participants will complete a 9-week, phone-based educational intervention that matches the PP intervention in terms of both time and attention.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Positive Psychology (PP) Intervention — This is an adapted, optimized, phone-based, 9-week positive psychology (PP) intervention. Participants will complete 9 weekly phone sessions (30 minutes each) with a study interventionist in which they will review PP exercises that they have independently completed in between phone sessions. The PP exercises will be completed in a treatment manual that describes the PP exercise and provides space to write about the exercise and its effects, and to answer associated questions. A total of 9 sessions will be completed over the course of the program.
  Arms: Positive Psychology (PP) Intervention
Behavioral: Educational Intervention — This is an educational intervention that will match the PP intervention in terms of both time and attention. Participants will complete 9 weekly phone sessions (30 minutes each) with a study interventionist in which they will review educational exercises that they have independently completed in between phone sessions. The exercises will be completed in a treatment manual that describes the exercise and provides space to write about the exercise and its effects, and to answer associated questions. A total of 9 sessions will be completed over the course of the program.
  Arms: Educational Intervention

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, preliminary effects, and candidate gut-brain mechanisms of an optimized positive psychology (PP) intervention for patients with irritable bowel syndrome (IBS), entitled "WISH," compared to an educational control intervention.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS), a disorder of gut-brain interaction (DGBI; also known as functional gastrointestinal (GI) disorder) is characterized by abdominal pain and altered bowel habits, and conceptualized as resulting from complex interactions between biological, psychological, and social factors. Compared to healthy populations, individuals with IBS have reduced positive psychological well-being, which in turn has been associated with impaired physical health, greater depression and anxiety, and worse health-related quality of life. A growing body of evidence supports the use of behavioral health interventions, referred to as brain-gut behavior therapies (BGBTs), as part of a comprehensive treatment approach for IBS. There is a critical need for new BGBTs for IBS that are scalable, acceptable, and mechanistically targeted.

Positive psychology (PP) interventions have successfully been implemented in a variety of other chronic medical conditions to improve well-being, health-related quality of life, health behavior engagement, and health outcomes. PP interventions are typically highly acceptable and easily delivered remotely without extensive specialized training, which increases their scalability and reach. Aside from the investigator's preliminary proof-of-concept work, however, PP interventions have not been evaluated in IBS.

Accordingly, the purpose of this study is to examine the feasibility, acceptability, preliminary eﬃcacy, and candidate gut-brain mechanisms of an optimized, 9-week, phone-delivered, PP intervention for patients with IBS, entitled "Well-being in IBS: Strengths and Happiness (WISH)," compared to a time-and attention-matched educational control intervention.

The primary aims of this randomized controlled trial (RCT) are to determine feasibility (at least 50% of participants completing at least 6/9 PP sessions) and acceptability (mean ease and utility ratings for each session of at least 7/10).

The exploratory aims of this RCT are to examine: (1) preliminary effects of the PP intervention in improving health-related (IBS symptom severity, health-related quality of life, and IBS diagnostic criteria), psychological (positive affect, optimism, resilience, self-eﬃcacy, depression, anxiety, GI symptom-specific anxiety, response to pain, and perceived stress), and health behavior (physical activity, avoidant/restrictive eating) outcomes; and (2) candidate gut-brain mechanisms of the PP intervention including changes in autonomic function (as measured by heart-rate variability), interoception, stress-mediated gene expression, and immune system activity.

ELIGIBILITY:
Inclusion Criteria:

* IBS Diagnosis: Adult patients with an IBS diagnosis meeting standardized Rome IV diagnostic criteria.
* Language and communication: English fluency and access to a phone.

Exclusion Criteria:

* Presence of inflammatory bowel disease or other structural/biochemical primary gastrointestinal illness that better explains IBS-like symptoms: As reported by the patient, their physician, and/or documented in the medical record.
* Severe psychiatric illness: Current manic episode, psychosis, or active substance use disorder diagnosed via the Mini International Neuropsychiatric Interview (MINI).
* Cognitive impairment: Assessed using a six-item cognitive screen developed for research.
* Presence of atrial fibrillation or a cardiac pacemaker, or daily use of beta blocking medication: As reported by the patient and/or documented in the medical record.
* Plans to start or participate in another new behavioral health intervention or psychotherapy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of Intervention Sessions Completed by Participants | Post-intervention at 9 weeks
  Feasibility will be measured by the proportion of intervention sessions completed by participants. The intervention will be considered feasible if at least 50% of participants complete at least 6/9 sessions.
Ease of Weekly Exercises | Weekly during intervention (weeks 1-8) and post-intervention (week 9)
  Participants will provide ratings of ease after each weekly exercise, measured on a 10-point Likert scale (0=very difficult, 10=very easy).
Utility of Weekly Exercises | Weekly during intervention (weeks 1-8) and post-intervention (week 9)
  Participants will provide ratings of utility after each weekly exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful).

SECONDARY OUTCOMES:
Immediate Impact of the Exercises: Change in Optimism Ratings | Weeks 1-9
  Participants will provide ratings of optimism before and after each positive psychology exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate higher levels of optimism.
Immediate Impact of the Exercises: Change in Happiness Ratings | Weeks 1-9
  Participants will provide ratings of happiness before and after each positive psychology exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate higher levels of happiness.
Immediate Impact of the Exercises: Change in IBS Knowledge Ratings | Weeks 1-9
  Participants will provide ratings of knowledge about IBS before and after each educational exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate higher levels of knowledge.
Change in IBS Symptom Severity | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the IBS symptom severity score (IBS-SSS) (Range 0-500). This is a validated disease-specific instrument that measures IBS symptom severity. Higher scores indicate more severe symptoms.
Change in IBS Health-Related Quality of Life | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the IBS Quality of Life (IBS-QOL) score (Range: 0-100), a validated disease-specific instrument measuring quality of life. Higher scores indicate better IBS-specific quality of life.
Change in Rome IV Diagnostic Criteria for IBS | At prescreening (prior to baseline), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the The Rome-IV Diagnostic Questionnaire - IBS Module, which is a validated disease-specific instrument used to screen for IBS diagnostic criteria and to provide a provisional (yes/no) diagnosis of IBS. To meet criteria for IBS, the following are required for the past 3 months: (1) recurrent abdominal pain at least weekly; (2) pain associated with 2 or more of the following criteria: a) related to defecation at least 30% of occasions; b) associated with change in stool frequency at least 30% of occasions; c) associated with change in stool form at least 30% of occasions; and (3) symptom onset at least 6 months prior to diagnosis.
Change in Positive Affect | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured with the positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses (Range: 10-50). Higher scores indicate higher levels of positive affect.
Change in Dispositional Optimism | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured with the Life Orientation Test-Revised (LOT-R), a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism.
Change in State Optimism | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured with the Brief State Optimism Measure (B-SOM), a validated 2-item instrument used to measure state optimism (Range: 0-100 for each item). Higher scores indicate greater state optimism.
Change in Resilience | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Brief Resilience Scale (BRS) (Range: 6-30), a reliable 6-item measure of the ability to "bounce back" or recover from stress. Higher scores reflect greater bounce back resilience.
Change in Self-Efficacy | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the General Self-Efficacy (GSE) Scale (Range: 10-40), a 10-item validated measure of self-efficacy, defined as an individual's perception of their ability to succeed at a task or achieve a goal. Higher scores indicate greater self-efficacy.
Change in Depression | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Hospital Anxiety and Depression Scale (HADS)-depression subscale. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
Change in Anxiety | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Hospital Anxiety and Depression Scale (HADS)-anxiety subscale. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
Change in Gastrointestinal (GI) Symptom-Specific Anxiety | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Visceral Sensitivity Index (VSI) score, a validated self-report measure of anxiety specific to visceral sensations (Range: 0-75). Higher scores indicate higher levels of GI-specific anxiety.
Change in Response to Pain | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Pain Catastrophizing Scale (PCS), a widely used tool to assess cognitive and affective responses to pain (Range: 0-52). Higher scores indicate higher levels of pain-related anxiety.
Change in Perceived Stress | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Perceived Stress Scale (PSS) (Range: 0-40), a validated measure to assess perceived levels of stress. Higher scores indicate higher perceived stress.
Change in Self-Reported Physical Activity | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the self-report International Physical Activity Questionnaire (IPAQ) Short Form. This 7-item measure assesses self-reported physical activity from the preceding 7 days. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. Higher scores reflect higher levels of physical activity.
Change in Avoidant and Restrictive Eating | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  Measured by the Nine Item Avoidant/Restrictive Food Intake Disorder screen (NIAS) (Range: 0-45), a validated tool to assess avoidant/restrictive eating patterns. Higher scores indicate higher levels of avoidant/restrictive eating patterns.
Change in Interoception | At baseline (week 1), at the mid-point of the intervention (week 5), post-intervention (week 9), and 3-months post-intervention (week 21)
  The Multidimensional Assessment of Interoceptive Awareness-Version 2 (MAIA-2) is a validated measure of interoception, defined as an awareness of internal bodily sensations (Range: 0-185). Higher scores indicate a higher level of interoceptive bodily awareness.
Change in Autonomic Function | At baseline (week 1) and post-intervention (week 9)
  Heart-rate variability measurements will be collected to explore changes in autonomic function related to the intervention.
Change in Stress-Mediated Gene Expression | At baseline (week 1) and post-intervention (week 9)
  Whole transcriptome analysis of blood samples by RNA sequencing (RNA-seq) will be completed to explore gene expression changes related to the intervention.
Change in Serum Cytokine Levels | At baseline (week 1) and post-intervention (week 9)
  Serum cytokine levels will be assessed to explore changes in immune system activity related to the intervention.
Treatment Credibility | Week 1 (after first phone session)
  The Credibility sub-scale (Range: 3-27) of the Credibility/Expectancy Questionnaire (CEQ) will be used to compare treatment credibility between conditions. Higher scores indicate higher treatment credibility.
Treatment Expectancy | Week 1 (after first phone session)
  The Expectancy sub-scale (Range: 3-27) of the Credibility/Expectancy Questionnaire (CEQ) will be used to compare treatment expectancy between conditions. Higher scores indicate higher treatment expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth N Madva, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To help advance other research, de-identified data will be shared via respective repositories as specified below:
  * Clinical data including demographics, self-report questionnaires, and heart-rate variability will be shared via the Vivli repository.
  * Genomic data generated from RNA-seq will be submitted as FASTQ files to the Database of Genotypes and Phenotypes (dbGaP) which will then be shared to the Sequence Read Archive (SRA) with controlled access.
Supporting Information: Study Protocol, SAP
Time Frame: Datasets will be provided to respective repositories by the end of the funding period. The clinical data shared with the Vivli repository will be archived and available for request by researchers for a minimum of 10 years after contribution. Genomic data will be preserved in the dbGaP/SRA repositories for at least three years following the completion of the grant.
Access Criteria: Clinical and genomic data will be shared with controlled access with the Vivli repository and dbGaP/SRA, respectively, for general research use, as allowed by the participants' informed consents and the Institutional Certification. Access to data requires the completion of a Data Use Agreement (DUA), which prohibits any redistribution or attempts to re-identify research participants.